CLINICAL TRIAL: NCT04678362
Title: TALazoparib and Avelumab as Maintenance Therapy in Platinum-Sensitive Metastatic or Locally Advanced URothelial Carcinoma: A Single-arm Phase 2 Trial
Brief Title: TALazoparib and Avelumab as Maintenance Therapy in Platinum-Sensitive Metastatic or Locally Advanced URothelial Carcinoma
Acronym: TALASUR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001105-24
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — talazoparib; avelumab

STUDY DESIGN:
Intervention Model Description: Single-arm phase 2 trial
Masking Description: None (open label=)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talazoparib+avelumab (Experimental): * Talazoparib will be administered at the daily dose of 1 mg given orally in a 28-day cycle, except for patients with mild renal impairment (Creatinine clearance 30-59 mL/min) who will receive 0.75 mg per day.
  * Avelumab will be administered by intravenous (I.V.) route over 60 minutes at the dose of 800 mg on D1 and D15, in a 28-day cycle.
  Interventions: Drug: Talazoparib + Avelumab

INTERVENTIONS:
Drug: Talazoparib + Avelumab — Patients will receive the combined treatment until the investigator considers that the patient no longer obtains benefit from it. The treatment will be continued until disease progression, unacceptable toxicity or discontinuation for any cause.

SUMMARY:
The main objectif is to determine the efficacy of a maintenance treatment combining Talazoparib and Avelumab after platinum-based chemotherapy in patients with locally advanced/metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
The first line treatment of urothelial carcinoma is a platinum-based chemotherapy. This treatment is efficient with a response rate > 50 % but the progression-free survival is short (7.7 months) and the chemotherapy is too toxic to be used in a prolonged time. Traditionally, maintenance chemotherapy refers to the utilization of regimens with less toxicity after the initial upfront treatment. This concept has already been efficient with PARP inhibitors in ovarian carcinoma and more recently with durvalumab in lung carcinoma.

The prevalence of somatic mutations in homologous recombination genes in UC as well as their association with platinum sensitivity suggests Talazoparib to be a target for a maintenance treatment of urothelial carcinoma. Moreover, there is a strong rational with both pre-clinical and clinical data to associate Avelumab and Talazoparib. This appears all the more relevant that Avelumab has already demonstrated its efficacy in urothelial carcinoma (after platinum-based chemotherapy failure).

In this context, the sponsorpropose a phase 2 study to assess the antitumor activity of the combination of Avelumab plus Talazoparib in metastatic urothelial carcinoma in maintenance therapy after platinum-based chemotherapy.

Considering the doubts about the best molecular predictive factors of Talazoparib and Avelumab, the sponsor willingly propose a non-selective study, without molecular screening. Tumors will be selected according to the platinum sensitivity which has the advantage to exclude poor prognosis tumors and will allow increasing the HRD tumor population.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years at the day of consenting to the study
* Provision of informed consent prior to any study specific procedures
* Histologically confirmed diagnosis of urothelial carcinoma of the renal pelvis, ureter (upper urinary tract), bladder or urethra. Both transitional cell and mixed transitional/non-transitional cell histologies are allowed, but transitional cell carcinoma must be the predominant histology.
* Documented Stage IV disease (T4b, N0, M0; any T, N1-N3, M0; any T, any N, M1) not candidate to a curative treatment with surgery or radiotherapy at the start of first-line platinum-based chemotherapy.
* Patient must have completed prior to inclusion a platinum-based (cisplatin or carboplatin) polychemotherapy for at least 4 cycles of chemotherapy (until 6 cycles maximum) and have a stable disease or a partial response (PR) or a complete response (CR) from the chemotherapy according to RECIST 1.1 criteria

  * A minimum dose of 55 mg/m² of cisplatin is required in order to count for 1 cycle.
* A minimum dose of carboplatin AUC 4.5 is required in order to count for 1 cycle
* Eligibility based on this criterion will be established locally by the investigator by examining pre and post-chemotherapy radiological assessments (CT/MRI)
* Neoadjuvant or adjuvant chemotherapy is allowed (with a delay of at least 12 months between the last dose of neoadjuvant or adjuvant chemotherapy and the relapse)
* Patient must be enrolled within 8 weeks after the last dose of chemotherapy and should start study treatment at least 3 weeks after the last dose of chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Hemoglobin ≥ 10.0 g/dL (patient may have been transfused before inclusion)
* Absolute neutrophil count (ANC) ≥1.5 x 109/L
* Platelet count ≥100 G/l
* Total bilirubin ≤1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤2.5 x ULN unless liver metastases are present in which case they must be ≤5x ULN
* Patient must have creatinine clearance estimated using the CKD equation of ≥ 40 mL/min
* Able to swallow and retain oral drug
* Life expectancy > 12 weeks
* Serum pregnancy test (for females of childbearing potential) negative at screening
* Male patient able to father children and female patient of childbearing potential and at risk for pregnancy must agree to use 2 highly effective methods of contraception throughout the study and for at least 60 days after the last dose of treatments
* Patient affiliated to a French Social Security System or a beneficiary of such a system
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
* Optional: provision of a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block (or subsection thereof) from the most recent primary or metastatic tumor biopsy

Exclusion Criteria:

* Patient who has never received chemotherapy with a platinum salt (cisplatin or carboplatin) for advanced/metastatic urothelial carcinoma
* Patient who has previously received more than one line of chemotherapy for advanced/metastatic urothelial carcinoma
* Patient whose disease has progressed according to RECIST v1.1 criteria after the first line platinum-based chemotherapy for urothelial carcinoma. The cancer must not be in the progression phase at inclusion
* Patient with known CNS metastases and/or carcinomatous meningitis
* Other malignancy within the last 3 years except: adequately treated non-melanoma, skin cancer curatively treated, in situ cancer of the cervix, ductal carcinoma in situ (DCIS), localized prostate carcinoma without PSA relapse
* Patient with myelodysplastic syndrome/acute myeloid leukemia history or with features suggestive of MDS/AML
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patient with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are allowed.Current treatment with an immunosuppressant medicinal product or treatment within 7 days prior to inclusion, EXCEPT:

  * Intra-nasal, inhaled or local steroids or local steroid injections (such as intra-articular injections)
  * Systemic corticosteroids at physiological doses of ≤ 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (such as CT scan premedication)
* Major surgery within 4 weeks or major radiotherapy within to starting experimental treatment. Previous palliative radiotherapy (≤ 10 fractions) for metastatic lesions is permitted provided that this has been completed at least one week prior to starting Talazoparib and Avelumab
* Active viral infection (HIV, Hepatitis B/C) or known history of positive test for HIV
* Any previous treatment with PARP inhibitor or any immunotherapy (e.g. anti-CTLA-4 or anti-PDL1/ PD1)
* Concomitant treatment with any drug on the prohibited medication list such as live vaccines, concomitant use of strong P-gp inhibitors (cf section "Prohibited concomitant treatments") or systemic corticoids at dose > 10 mg/day prednisone or equivalent. Live vaccines administered more than 30 days before study entry are permitted
* Clinically significant (e.g. active) cardiovascular disease cerebral vascular accident/stroke in the 3 months prior to enrollment: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure (≥ New York Heart Association Classification Class II), serious cardiac arrhythmia requiring medication, uncontrolled high blood pressure, cerebrovascular accident, transient ischaemic attack
* Patient considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease or any psychiatric disorder that prohibits obtaining informed consent
* Pulmonary embolism or deep vein thrombosis within 3 months prior to inclusion (unless if stable, asymptomatic and treated with a low molecular heparin for at least 10 days prior to starting Talazoparib + Avelumab).
* Pregnant or lactating woman;
* Participation in another interventional study with a systemic anti-cancer treatment within 4 weeks prior to inclusion. Inclusion in observational or interventional studies not involving a health product is permitted. Patient with telephone follow up of toxicities and simple laboratory monitoring or other questionnaires alone may be included.
* Patient unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication;Previous organ transplant including stem cell allotransplantation or double umbilical cord blood transplantation.
* Patient with a known hypersensitivity to Talazoparib and Avelumab or any of the excipients of the product.
* People who are vulnerable under the law (minors, adults under legal protection, people deprived of their freedom)
* Other persisting toxicities related to previous anticancer treatments: "Persisting toxicity related to prior therapy (NCI CTCAE Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival | 7 months

SECONDARY OUTCOMES:
Overall Survival | 18 months
Duration of tumoral response | 18 months

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU Jean Minjoz, Besançon
  - Centre François baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George-François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hospices civils de Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - Croix Saint-Simon Diaconesses, Paris
  - Hopital Tenon, Paris
  - Centre Eugène Marquis, Rennes
  - IUCT, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coquan E, Clarisse B, Lequesne J, Brachet PE, Neviere Z, Meriaux E, Bonnet I, Castera M, Goardon N, Boutrois J, Travers R, Joly F, Grellard JM, Thiery-Vuillemin A. TALASUR trial: a single arm phase II trial assessing efficacy and safety of TALazoparib and Avelumab as maintenance therapy in platinum-Sensitive metastatic or locally advanced URothelial carcinoma. BMC Cancer. 2022 Nov 24;22(1):1213. doi: 10.1186/s12885-022-10216-z. PMID 36434554